CLINICAL TRIAL: NCT01503177
Title: A Phase 1 Trial of Oncolytic Measles Virotherapy in Mesothelioma
Brief Title: Intrapleural Measles Virus Therapy in Patients With Malignant Pleural Mesothelioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1023; NCI-2011-03574 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-12-16; First posted 2012-01-02 (Estimated); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Recurrent Malignant Mesothelioma; Stage IA Malignant Mesothelioma; Stage IB Malignant Mesothelioma; Stage II Malignant Mesothelioma; Stage III Malignant Mesothelioma; Stage IV Malignant Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Photons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (viral therapy) (Experimental): Patients receive MV-NIS intrapleurally on day 1. Treatment repeats every 28 days for up to 6 courses in absence of disease progression or unacceptable toxicity.
  Interventions: Biological: oncolytic measles virus encoding thyroidal sodium iodide symporter; Other: laboratory biomarker analysis; Procedure: single photon emission computed tomography; Procedure: computed tomography

INTERVENTIONS:
Biological: oncolytic measles virus encoding thyroidal sodium iodide symporter — Given intrapleurally
  Other Names: MV-NIS
Other: laboratory biomarker analysis — Correlative studies
Procedure: single photon emission computed tomography — Correlative studies
  Other Names: SPECT imaging; tomography, emission computed, single photon
Procedure: computed tomography — Correlative studies
  Other Names: tomography, computed

SUMMARY:
This phase I clinical trial investigates the side effects and the best dose of local (intrapleural measles virus therapy in treating patients with malignant pleural mesothelioma (MPM). The investigators anticipate that the intrapleural of the vaccine strain measles virus will enable the virus to specifically infect and kill cancer cells and spare, without damaging normal cells. Furthermore, the investigators expect the measles virus to trigger an anti-tumor immune response which will result in additional destruction of the tumor by immune cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Maximum tolerated dose (MTD) for the intrapleural administration of a modified vaccine strain measles virus (MV) genetically engineered to produce human thyroidal sodium iodine symporter (NIS) (MV-NIS [oncolytic measles virus encoding thyroidal sodium iodide symporter])in patients with MPM.

SECONDARY OBJECTIVES:

Safety and toxicity of the repeated (up to 6 cycles) intrapleural administration of MV-NIS in patients with malignant pleural mesothelioma.

TERTIARY OBJECTIVES:

I. Time course of viral infection, dissemination and elimination by non-invasive measurements of NIS gene expression using radioactive iodine and single-photon emission computed tomography (SPECT)/ computed tomography (CT) imaging with.

II. Viremia, viral replication, and viral shedding following intrapleural administration.

III. Changes in humoral and cellular anti-MV immunity following the intrapleural administration of MV-NIS.

IV. Antitumor efficacy of this approach by serial measurements of radioiodine uptake by SPECT/CT, radiographic response, and time to disease progression.

V. Changes in both local and systemic innate and adaptive anti-tumor immunity following the intrapleural administration of MV-NIS.

VI. Effect of MV-NIS administration on the eukaryotic initiation factor (eIF) 4F translation complex in mesothelioma cells.

OUTLINE: This is a dose-escalation study.

Patients receive the oncolytic measles virus encoding thyroidal sodium iodide symporter (MV-NIS) intrapleurally. In the absence of unacceptable side effects or disease progression treatment can be repeated every 28 days for up to 6 courses.

After completion of study treatment, patients are followed up every 3 to 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

PRE-REGISTRATION:

* Diagnosis of MPM, confined to single pleural cavity, with histologic confirmation of the primary tumor
* Measurable disease per modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria for mesothelioma
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0, 1, or 2
* Ability to provide informed consent
* Willingness to return to Mayo Clinic Rochester or the University of Minnesota Cancer Center for follow up
* Life expectancy >= 12 weeks (in the opinion of the enrolling investigator)
* Willingness to provide the biologic specimens and participate in the SPECT/CT imaging as required by the protocol
* Presence of a pleural effusion with the ability to safely place an intrapleural catheter or have pre-existing intrapleural catheter
* Absolute neutrophil count (ANC) >= 1500/μL
* Platelet count >= 100,000/μL
* Total bilirubin =< 1.5 x upper limit of institutional normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 2 x upper limit of institutional normal
* Serum Creatinine =< 1.5 x upper limit of institutional normal
* Hemoglobin >= 9.0 g/dL
* Must be willing to implement contraception throughout study and for the 4 weeks following last viral administration

REGISTRATION:

* Anti-measles immunity as demonstrated by serum IgG anti-measles antibody levels of ≥ 1.1 EU/ml as determined by BioPlex Measles IgG multiplex flow immunoassay.
* Hepatitis B and C negative
* Human immunodeficiency virus (HIV) negative
* CD4 count >= 200/μL
* CT imaging review submission to confirm unilateral pleural involvement; this review for CT imaging is mandatory prior to registration to confirm eligibility; it should be initiated as soon as possible after pre-registration
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only

Exclusion Criteria:

PRE-REGISTRATION

* Uncontrolled intercurrent illness including, but not limited to:

  * Active infection =< 5 days prior to pre-registration
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Symptomatic congestive heart failure New York Heart Association classification III or IV
  * Symptomatic coronary artery disease (CAD)
  * Symptoms of CAD on systems review
  * Cardiac arrhythmias

Any of the following therapies prior to pre-registration:

* Chemotherapy =< 4 weeks
* Immunotherapy =< 4 weeks
* Biologic therapy =< 4 weeks; Note exception: prior viral and/or gene therapy are exclusion criteria
* Radiotherapy =< 4 weeks Failure to fully recover from acute, reversible effects of prior anti-cancer therapy regardless of interval since last treatment; NOTE: patients must have fully recovered from all acute, reversible toxicities (defined as Common Terminology Criteria for Adverse Events [CTCAE] 4.0 =< grade 1) associated with previous treatment

Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

* Pregnant women
* Nursing women
* Men or women of childbearing potential who are unwilling to employ adequate contraception

  * Any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA] approved indication and in the context of a research investigation) or any other treatment specifically for treating the current malignancy
  * Immunocompromised patients, including patients known to be HIV positive
  * Other active malignancy =< 2 years prior to pre-registration; EXCEPTIONS: non-melanotic skin cancer or carcinoma-in-situ of the cervix
  * History of organ transplantation
  * Known hepatitis B or C
  * Treatment with oral/systemic corticosteroids; NOTE: with the exception of topical or inhaled steroids
  * Exposure to household contacts =<15 months old or household contact with a person with known immunodeficiency
  * Allergy to measles vaccine or history of severe reaction to prior measles vaccination
  * Allergy to iodine; NOTE: this does not include reactions to intravenous contrast materials
  * History of tuberculosis or purified protein derivative (PPD) skin test positivity
  * Inability or unwillingness to have pleural catheter placed
  * Requiring ongoing blood product support at time of pre-registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-11 (Actual)

PRIMARY OUTCOMES:
Adverse event (AE) profile | 90 Days
  The number and severity of toxicity incidents will indicate the level of tolerance for MV-NIS in the therapy of MPM. Non-hematologic toxicities will be evaluated via the CTCAE v4.0 standard toxicity grading. Hematologic toxicity measures such as anemia, neutropenia and thrombocytopenia will be assessed using continuous variables as the outcome measures (nadir and percent change from baseline values) as well as categorization via CTCAE v4.0 standard toxicity grading. Frequency distributions and other descriptive measures will form the basis of the analysis of these variables.

SECONDARY OUTCOMES:
Describe the safety of the intrapleural administration of MV-NIS in patients with malignant pleural mesothelioma for all cycles out to 90 days. | 90 Days
  The number and severity of adverse events (AE) over the course of up to 6 cycles of MV-NIS therapy will indicate the level of tolerance for MV-NIS in the therapy of MPM. AE will be evaluated similar to the primary outcome via the CTCAE v4.0 standard toxicity grading and frequency distributions and other descriptive measures will form the basis of the analysis of these variables.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Peikert, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States